CLINICAL TRIAL: NCT04147312
Title: The Study on the Clinical Value of Fufang E'Jiao Jiang Intervening Cancer-related Fatigue (Deficiency of Qi and Blood)
Brief Title: Fufang E'Jiao Jiang Intervening Cancer-related Fatigue
Acronym: FFEJJICRF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); Shandong University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2018YFC1707406
Record Dates: First submitted 2019-09-01; First posted 2019-11-01 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2019-08

CONDITIONS: Cancer-related Fatigue
Keywords: Traditional Chinese medicine; Fufang E'Jiao Jiang; Randomized controlled trial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Fufang E'Jiao Jiang, 20milliliters(mL) once, 3 times a day, continuous intervention for 21days each cycle, and use 2 cycles
  Interventions: Drug: Fufang E'Jiao Jiang
- control group (Placebo Comparator): Placebo containing low-dose Fufang E'Jiao Jiang, 20mL once, 3 times a day, continuous intervention for 21 days each cycle, and use 2 cycles
  Interventions: Drug: placebo containing low-dose fufang E'Jiao Jiang

INTERVENTIONS:
Drug: Fufang E'Jiao Jiang — Fufang E'Jiao Jiang, 20milliliters(mL) once, 3 times a day, continuous intervention for 21 days each cycle, and use 2 cycles
  Other Names: A listed Chinese Medicine
  Arms: Treatment group
Drug: placebo containing low-dose fufang E'Jiao Jiang — placebo containing low-dose Fufang E'Jiao Jiang, 20mL once, 3 times a day, continuous intervention for 21 days each cycle, and use 2 cycles
  Other Names: placebo
  Arms: control group

SUMMARY:
With the therapeutic tool of carcinoma increasing, life span extending, the solicitude for the patients'quality of life appear more important. Cancer-related fatigue (CRF) is one of the most prevalent and debilitating symptoms experienced by people with cancer. It can persist for months or years after cancer therapy is completed and has a negative impact on all areas of function. Meaningful evidence-based treatment options for CRF are extremely limited and finding safe, inexpensive, and effective interventions for managing this distressing symptom are urgently needed. Our previous clinical experience have shown that traditional Chinese medicine（TCM） had a great effect on improving CRF, Several studies proven that its'mechanism were related to the regulation of immune function and endocrine hormones. Fufang E'Jiao Jiang (FFEJJICRF) is a commonly-used Chinese patent medicine and successfully marketed in China for many years, which are effective in improvement for TCM symptoms of deficiency with qi and blood. This proposal will investigate the effects of FFEJJICRF on CRF among non-small cell lung cancer, colorectal cancer, and gastric cancer, so as to find a new way for curing it in clinical.

DETAILED DESCRIPTION:
By conducting large sample, multicenter, double-blind, randomized comparison clinical research, this test will investigate the effects of fufang E'Jiao Jiang intervening cancer-related fatigue (CRF) with deficiency of qi and blood, under the guidance of its specification. This test choose the improvement of fatigue degree as key indicator, and choose the improvement both symptoms of patients and quality of life as second indicators. And last, the study will try to verify its safety and efficacy with some haematological indexs and reveal its mechanism from the perspectives of hormone, immune and metabonomics, so as to explore the advantages of traditional Chinese medicine（TCM） in the treatment of CRF and support some high quality, internationally recognized clinical evidence.

ELIGIBILITY:
Inclusion Criteria:

1. The age of patients between 18 and 75，gender not limited.
2. Patients that pathologically diagnosed with colorectal cancer, non-small cell lung cancer (NSCLC) or gastric cancer.
3. The patients' TNM stage of NSCLC is IIIB-IV, colorectal cancer is IV, and gastric cancer is IV, in addition all of them should be with tumors that can not be radically resected.
4. If patients have not received chemotherapy, they should be evaluated that tumor will not progress within 30 days, and their bodies can tolerate intravenous targeted therapy.
5. Patients who meet the diagnostic criterion for cancer related fatigue with deficiency of qi and blood.
6. The expected survival period is more than 3 months.
7. Fatigue score evaluated by visual analogue fatigue scale isn't lower than 4, and Karnofsky scale score isn't lower than 60.
8. Good compliance and agreeable to sign an informed consent before test.
9. Subjects agree not to participate in other intervention studies during test.

Exclusion Criteria:

1. Those who need immunotherapy or radiotherapy during the test.
2. Those who have significant trauma injuries in the past one month.
3. Those who have severe bleeding or systemic infection diseases that had not been completely controlled.
4. Those who have tangible proofs of marrow or central nervous system metastasis.
5. Those who have received erythropoietin or blood transfusion within 1 month before test.
6. Those who have hypersplenism, hyperthyroidism, desmosis, tuberculosis and other diseases that have not been completely controlled.
7. Those who complicated with serious diseases such as cardiovascular or cerebrovascular system diseases, active hepatitis, disfunction of liver or kidney.
8. Those who are known or suspected to be allergic to test drugs.
9. Those who have eaten EJiao products in the past 2 weeks.
10. Those who have occurred Ileus.
11. Those suffering from severe malabsorption or other diseases that affect gastrointestinal absorption.
12. Those who cannot understand, read and fill in the self-rating scale due to their level of knowledge or intelligence.
13. Those who may happen any unstable conditions or conditions that endanger the patient's safety or compliance, for example the spirits.
14. Those who have been diagnosed with other malignant tumors (except fully treated cervix and skin carcinoma in situ, or other tumors that have been surgically cured and not recurred for at least 5 years) .
15. Those who participated in other therapeutic clinical trials within 30 days.
16. Pregnant or nursing women, or childbearing female that are inadequate contraception.
17. Those who are inappropriate to participate in the study determined by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-10-17 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Fatigue degree with the Piper fatigue scale (Piper) | 6 weeks
  Piper is composed of 24 questions assessing total CRF, as well as subscales of behavioral, affective, sensory, and cognitive/mood fatigue. Each question is cored from 0 to10 points, where a higher score indicates severe symptoms; 1 to 3 point is mild, 4 to 6 point is moderate, and 7 to 10 point is severe. Piper is taken at the baseline, 1 weeks, 3 weeks,4 weeks, and 6 weeks after treatment

SECONDARY OUTCOMES:
The occurrence of myelosuppression during chemotherapy | 10 weeks
  1)the duration time of myelosuppression; 2) the proportion among them that should be intervened with salvage treatments; the salvage treatments, including their variety, quantity and duration times; 3) the incidence and duration time of grade 3-4 myelosuppression. Those measurements were recorded and calculated separately at the end of the study.
The amounts of leukocyte cells, hemoglobin and platelet in peripheral blood | 10 weeks
  Those who are receiving chemotherapy should be measured at the baseline, 1 weeks, 3 weeks,4 weeks, 6 weeks and 10 weeks after treatment. Those who are not receiving chemotherapy should be measured at the baseline, 3 weeks, 6 weeks, 10 weeks.
Change of patients' living quality with the Edmonton symptom assessment scale(ESAS) | 10 weeks
  Changes of patients' living quality with ESAS to measure participants'responses to 11 common symptoms (pain, fatigue, nausea, depression, anxiety, drowsiness, shortness of breath, appetite, sleep problems, feeling of well-being and pruritus). Intensity of symptoms rated on a 0 to 10 scale from 0 "no symptom" to 10 "worst possible symptom"
Change of patients' functional status with Karnofsky performance status (KPS) | 10 weeks
  KPS Scores ranged from 100 to 0,The higher score represent the better health, the more likely that you are able to tolerate the side effects of treatment. It is generally considered that Karnofsky80 score or above represent patients can live independently, 60~80 score represent semi-independently, Under 60 represent patients often need help in living.
Quality of Life with Functional assessment of cancer therapy-fatigue（FACT-F） | 6 weeks
  FACT-F investigates participants from six dimensions (physiology, social/family status, emotion, function, fatigue, tumor) and each question is rated on a 5-point Likert scale. Higher scores represent more agreeable with the content of the items
Aldosterone, insulin-like growth factor, cortisol, growth hormone | 6 weeks
  Levels of serum hormone on aldosterone, insulin-like growth factor, cortisol, growth hormone
Change from baseline in lymphocyte subsets counts up to 6 Weeks: T Cell, B Cell, Natural Killer Cell (T,B,NK) | 6 weeks
  Lymphocyte subsets include T cell, B cell and Natural killer (NK) cells
Change from baseline in T-cells Subsets Counts up to 6 Weeks: T-Cells Subsets | 6 weeks
  T-cells Subsets Counts up to 6 Weeks: T-Cells Subsets
T-Cell Cytokines | 6 weeks
  T-cell cytokine subsets include IFNγ, IL-1β,IL-2,IL-4,IL-5,IL-6,IL-8,IL-10,IL-12p70,IL-17A,IL-17F,IL-22,TNFα,TNFβ
Circulating metabolite concentrations by nontargeted metabolomics techniques | 6 weeks
  Blood concentrations of metabolites including amino acids, acylcarnitines, hexoses, biogenic amines, phosphatidylcholines, and sphingomyelins
Triiodothyronine, free triiodothyronine, bound thyroxine, free thyroxine, thyroid stimulating hormone | 6 weeks
  Thyroid hormones index

OTHER OUTCOMES:
Adverse reaction rates, including the damage of liver and renal functions that reflected by increased alanine aminotransferase, aspartate aminotransferase and creatinine urea nitrogen respectively | 6 weeks
  Safety evaluation
Percentage of patients who dropout by other adverse reactions caused by drugs | 6 weeks
  Another safety evaluation: Percentage of patients who dropout by other adverse reactions caused by drugs meanwhile excluding myelosuppression (grading standard of adverse reactions according to the evaluation standard of CTCAE v4.03)
Collect costs of the whole observation period, and count the cost-effectiveness analysis based on the outcome of clinical study | 6 weeks
  Evaluation of health economics

CONTACTS AND LOCATIONS:
Overall Officials: xu yun, doctor, Study Director — Xiyuan Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Oncology Department of Xiyuan hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Song Z, Sun LY, Gu SS, Zhu XS, Lai HZ, Lu F, Cui N, Li QY, Wu Y, Xu Y. Exploring the Safety, Effectiveness, and Cost-Effectiveness of a Chinese Patent Medicine (Fufang E'jiao Syrup) for Alleviating Cancer-Related Fatigue: A Protocol for a Randomized, Double-Blinded, Placebo-Controlled, Multicenter Trial. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211002919. doi: 10.1177/15347354211002919. PMID 33834863